CLINICAL TRIAL: NCT07380178
Title: The Effect of Apple Fruit Extract (Malus Sylvestris Mill) as an Antioxidant and Anti-Inflammatory on Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Niken Dyah Aryani Kuncorowati, Otolaryngologist (ENT Specialist), Universitas Sebelas Maret
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 007/12/2024
Record Dates: First submitted 2025-07-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: allergic rhinitis; quercetin; antioxidant; anti-inflammatory
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Quercetin; apple polyphenol extract; Loratadine; fluticasone furoate

STUDY DESIGN:
Intervention Model Description: 4 group study
Masking Description: Department Biomedic and Science Universitas Sebelas Maret Surakarta Indonesia, Department Pharmacy Universitas Muhammadiyah Surakarta Indonesia, Universitas Sebelas Maret Hospital Sukoharjo Indonesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Experimental): Loratadine 10 mg/day and Fluticasone Furoate 27.5 mcg twice daily.
  Interventions: Other: Loratadine 10 Mg; Other: Fluticasone Furoate
- Treatment A: Quercetin 100 mg (Experimental): Loratadine 10 mg/day, Fluticasone Furoate 27.5 mcg twice daily, and Quercetin 100 mg/day.
  Interventions: Other: Quercetin; Other: Loratadine 10 Mg; Other: Fluticasone Furoate
- High-Dose Quercetin (Experimental): Loratadine 10 mg/day, Fluticasone Furoate 27.5 mcg twice daily, and Quercetin 200 mg/day.
  Interventions: Other: Quercetin; Other: Loratadine 10 Mg; Other: Fluticasone Furoate
- Apple Extract Only (Experimental): Apple fruit extract (Malus sylvestris Mill) and Quercetin 200 mg/day.
  Interventions: Other: Quercetin; Other: Apple Extract

INTERVENTIONS:
Other: Quercetin — In the treatment group, standard therapy is given along with additional quercetin at different doses.
  Arms: Apple Extract Only; High-Dose Quercetin; Treatment A: Quercetin 100 mg
Other: Apple Extract — In the treatment group is give of Apple extract
  Arms: Apple Extract Only
Other: Loratadine 10 Mg — Control Loratadine 10 mg/day
  Arms: Control Group; High-Dose Quercetin; Treatment A: Quercetin 100 mg
Other: Fluticasone Furoate — Control Fluticasone Furoate 27.5 mcg twice daily
  Arms: Control Group; High-Dose Quercetin; Treatment A: Quercetin 100 mg

SUMMARY:
This study was conducted to see before and after treatment whether it provided improvement in the patient's clinical symptoms.

DETAILED DESCRIPTION:
This research is the first to be conducted with preliminary research on humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 60 years who have signed an informed consent
* Diagnosed with persistent allergic rhinitis with a Skin Prick Test or Positive IgE Examination.

Exclusion Criteria:

* The presence of complications in the nose such as nasal septum deviation, polyps, rhinosinusitis
* Have undergone specific immunotherapy for 2 years
* Use of drugs that affect allergy test results: antihistamines, corticosteroids, antihypertensive drugs, and decongestants
* Pregnancy and Breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — age 18 - 60 years
Enrollment: 40 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | Baseline, Month 3, and Month 6
  The TNSS evaluates the severity of four nasal symptoms: nasal congestion, sneezing, nasal itching, and rhinorrhea. Each symptom is rated on a 4-point scale: 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The total score is the sum of the four individual symptom scores, ranging from 0 to 12. Higher scores indicate worse symptom severity.

SECONDARY OUTCOMES:
Serum Interleukin-6 (IL-6) Levels | Baseline, Month 3, and Month 6
  Concentration of IL-6 measured using Enzyme-Linked Immunosorbent Assay (ELISA).
Malondialdehyde (MDA) Levels | Baseline, Month 3, and Month 6
  Oxidative stress marker measured using ELISA kit.
Nuclear Factor-Kappa Beta (NF-kB) Expression | Baseline, Month 3, and Month 6
  Transcription factor expression by ELISA assay.
Serum Interleukin-8 (IL-8) Levels | Baseline, Month 3, and Month 6
  Concentration of IL-6 measured using Enzyme-Linked Immunosorbent Assay (ELISA).
Serum TNF-alpha Levels | Baseline, Month 3, and Month 6
  Concentration of TNF-alpha measured using Enzyme-Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sebelas Maret Hospital, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
This research is related to the results of the dissertation as a requirement for graduating from a doctoral degree

REFERENCES:
- See also: protocol research — https://drive.google.com/drive/folders/1uqJgY9UBYk_AbJwBA8OokIoSUOFjSZc8?usp=drive_link
- Available data/document: Individual Participant Data Set: Niken Dyah Aryani K,MD,ORL-HNS — https://drive.google.com/drive/folders/12UPXOBkPG0U5BfQb_PVfP5v-INJWqSTx?usp=drive_link — Thank you and I hope this research can be used as a basis for additional therapy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT07380178/Prot_SAP_000.pdf